CLINICAL TRIAL: NCT06308237
Title: Effects of Resisted Versus Balance Exercises on Cognitive And Motor Function In Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0293
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Motor control; Randomized clinical trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (RESISTED EXERCISES) (Experimental): Group A will receive a session of resisted exercises for 30 minutes. Treatment session will be given for 3 days per week for 12 weeks. This resisted training exercise program consist of three phases: Warm-up phase (5 minutes, after Warm-Up phase 20 minutes resisted exercise training then cooling phase (5 minutes).
  Interventions: Other: RESISTED EXERCISES
- GROUP B (BALANCE EXERCISES) (Experimental): Group B will receive a session of Balance exercises for 30 minutes. Treatment session will be given for 3 days per week for 12 weeks. This balance exercise program consist of three phases:Warm-up phase (5 minutes), after Warm-Up phase, 20 minutes balance exercise training then cooling phase (5 minutes).
  Interventions: Other: BALANCE EXERCISES

INTERVENTIONS:
Other: RESISTED EXERCISES — Patients will perform Chest plank for 30 seconds with 4 repetitions.
  Then the Participants will perform these exercises for 1 minute each with 4 repetitions:
  Wide grip lateral pull down , Lying triceps press, Sit up squats, Barbell curl each.
  And will perform Thigh adduction for1 minute with 2 repititions.
  Arms: GROUP A (RESISTED EXERCISES)
Other: BALANCE EXERCISES — Static and dynamic balance exercises will include:
  Patients will perform Arm abduction holding a half-kg dumbbell, Opposite arm and leg in a quadruped position, Walking in a tandem stance(forward and backward), Turning and bending to the sides in a standing position, Pass through obstacles in a spiral, for 2 minutes each.
  Then they will perform throwing a medicine ball to investigator and back while trying to maintain balance, Tandem stance, Walking backwards, Two-leg bridge as well as single (2 repetitions), Leg bridge (raising the other leg), walking on the heel, performing rhythmic movements while stepping on a circular environment and balance board exercises, for 1 minute each.
  And will Walk up and down the stairs for 3 minutes.
  Arms: GROUP B (BALANCE EXERCISES)

SUMMARY:
Mild cognitive impairment affects older adults and it includes memory and attentions deficits, and problem-solving difficulties in activities of daily living. Resisted exercises is considered a viable strategy to improve balance and motor function in older population. Balance exercises comprises proprioceptive, visual and motor learning to a larger degree and has positive effects on memory and spatial cognition and improves balance and motor function. This study aims to determine the effects of resisted and balance exercises on cognition and motor function in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Aziz Bhatti Shaheed Teaching Hospital Gujrat in seven months after approval of synopsis. The sample size for this trial is 78 patients with MCI. The participants will be randomly allocated into two groups using Online Randomization tool. Group A will receive resisted exercises for 30 minutes and Group B will receive balance exercises for 30 minutes. Participants will receive 3 sessions on alternate days per week for 12 weeks.Montreal Cognitive Assessment (MoCA) and Computerized battery test will be used to assess cognitive impairment, Mini-besTest and Time Up and Go Test (TUG) for balance and motor function.Data will be entered and analysed by using SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Mild Cognitive Impairment. (Having score between 18 - 24) on MoCA.
2. Participants with Both Genders will be included .
3. The Age limit for the participants will be 60 to 75 years.
4. Patients having Independence of life (ability to walk independently without any walking aid).

Exclusion Criteria:

1. Previous and current History Cardiovascular, neurological, psychiatric and motor disorders like (fractures, diagnosis of Osteoporosis)
2. Patients taking any medication for mild cognition.
3. Depressive symptoms, acute and chronic conditions that would preclude exercise, regular exercise (>30 min/day, >3days/week).
4. Patients having estrogen replacement therapy.
5. Simultaneous participation in other studies.
6. Regular physical activity (once a week during the last 3 months); physio therapeutic treatment in the last 3 months.
7. Diseases that promote incapacity; severe visual deficiency; recurrent vertigo; and uncontrolled systemic arterial hypertension.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
MoCA (Montreal Cognitive Assessment ) | 14th week
  The Montreal Cognitive Assessment (MoCA) will be used as a screening tool as well as assessment tool for cognition. It is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer
Mini-Balance Evaluation Systems Test (BESTest). | 16th week
  It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits.It is a 14-item test scored on a 3-level ordinal scale.
Timed UP and GO Test (TUG) : | 16th week
  The Timed Up and Go test (TUG) will be used as a screening as well as assessment scale for balance and motor function. It can measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.This test has been used extensively in geriatric medicine to examine balance, gait speed, and functional ability that would be required for the performance of basic activities of daily living in older people.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Phd-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No